CLINICAL TRIAL: NCT06657261
Title: Comparison of the Analgesic Efficacy of Deep and Superficial Serratus Anterior Plane Block With the Combination of Deep Serratus Anterior Plane and Transverse Thoracic Muscle Plane Block in Coronary Artery Bypass Surgery: A Randomized Controlled Trial
Brief Title: Comparison of the Analgesic Efficacy of Chest Wall Blocks in Coronary Artery Bypass Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AsenaIremYildiz2
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Arterial Disease (CAD); Serratus Anterior Muscle Plane Block; Transversus Thoracis Muscle Plane Block; Postoperative Analgesia

STUDY DESIGN:
Intervention Model Description: "The anesthesia and surgical method will be the same for both patient groups. One group of patients will receive deep and superficial serratus anterior plane block. The other group will receive a combination of deep serratus anterior plane block and transverse thoracic muscle plane block. Postoperative visual pain scores will be observed for both groups. At the end of the study, the analgesic efficacy of the two groups will be compared."
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The patient group receiving deep and superficial serratus anterior plane block (Active Comparator): In this group, the ultrasound probe will be placed on the 5th rib in the mid-axillary line. After visualizing the muscle structures down to the rib (latissimus dorsi, teres major, and serratus anterior), the needle will be advanced using the in-plane technique to two separate areas on the 5th rib: the superficial and deep fascial planes of the serratus anterior muscle. A total of 20 ml of 0.25% bupivacaine will be injected into both areas. The procedure will be performed bilaterally.
  Interventions: Procedure: The patient group receiving deep and superficial serratus anterior plane block
- The patient group receiving a combination of deep serratus anterior plane block and transverse thora (Active Comparator): In this group, for the TTMP block, the ultrasound probe will be placed on the midclavicular line at the 3rd or 4th intercostal space, where the pleura, pectoralis major, and intercostal muscles will be visualized. A lateral-to-medial scan will be performed to visualize the hypoechoic TTMP located deep to the intercostal muscle and above the pleura. The needle target will be the plane between the internal intercostal muscle and the TTMP. In this area, 10 ml of 0.25% bupivacaine will be injected. The procedure will be performed bilaterally. For the deep SAPB, the ultrasound probe will be placed on the 5th rib in the mid-axillary line. After visualizing the muscle structures down to the rib (latissimus dorsi, teres major, and serratus anterior), the needle will be advanced using the in-plane technique to the fascial plane deep to the serratus anterior muscle on the 5th rib. In this area, 10 ml of 0.25% bupivacaine will be injected. The procedure will be performed bilaterally.
  Interventions: Procedure: The patient group receiving a combination of deep serratus anterior plane block and transverse thoracic muscle plane block

INTERVENTIONS:
Procedure: The patient group receiving deep and superficial serratus anterior plane block — The ultrasound device to be used , the type of single-use ultrasound-compatible block needle, the type of local anesthetic agent to be administered to the patient, the concentration of the local anesthetic agent, and the total dose of the local anesthetic agent to be administered to the patient will be the same.
  Arms: The patient group receiving deep and superficial serratus anterior plane block
Procedure: The patient group receiving a combination of deep serratus anterior plane block and transverse thoracic muscle plane block — The ultrasound device to be used , the type of single-use ultrasound-compatible block needle, the type of local anesthetic agent to be administered to the patient, the concentration of the local anesthetic agent, and the total dose of the local anesthetic agent to be administered to the patient will be the same.
  Arms: The patient group receiving a combination of deep serratus anterior plane block and transverse thora

SUMMARY:
In this study, the analgesic effects of the Transverse Thoracic Muscle Plane Block and deep Serratus Anterior Plane versus deep and superficial Serratus Anterior Plane applications, which will be performed under ultrasound guidance in patients undergoing coronary artery bypass surgery with sternotomy, will be compared and evaluated.

DETAILED DESCRIPTION:
Postoperative pain is a critical risk factor for the development of pulmonary and cardiovascular complications in coronary artery bypass graft (CABG) surgery. If effective respiratory function cannot be maintained in patients with high pain levels, atelectasis, cardiac ischemia, and arrhythmias may be observed. This prolongs the hospital discharge time of patients and increases the frequency of postoperative pulmonary complications and postoperative morbidity. Moreover, if postoperative acute pain is not adequately treated, chronic pain may develop after surgery, preventing patients from regaining their normal activities for a long time. In addition to medications, various neuroaxial and peripheral nerve blocks can be used in cardiac surgery. The use of intraoperative heparin limits the application of neuroaxial anesthesia (thoracic epidural and intrathecal opioids) and paravertebral block due to potential complications. Nevertheless, studies have shown their benefits in reducing cardiac and pulmonary complications. Recently, fascial plane nerve blocks, which are alternatives to these methods, have gained more popularity in cardiovascular surgery. These blocks include pectoral nerve blocks, serratus anterior plane block (SAPB), erector spinae plane block (ESPB), transverse thoracic plane blocks (TTMP), pecto-intercostal fascial blocks (PIF), and intercostal nerve blocks. The inability to effectively prevent postoperative pain in cardiac surgery has led not only to the exploration of new block applications but also to the combination of these blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80
* Patients with ASA score I-II-III
* Patients with a body mass index (BMI) between 18-35
* Patients undergoing sternotomy in the operating room

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* Patients with an ASA score of IV or higher
* Patients with advanced comorbidities
* Patients with a history of bleeding diathesis
* Patients using medications that cause bleeding disorders
* Patients with infections in the area where the block will be performed
* Patients with a body mass index (BMI) below 18 or above 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Analgesic Efficacy of Deep and Superficial Serratus Anterior Plane Block with the Combination of Deep Serratus Anterior Plane and Transverse Thoracic Muscle Plane Block in Coronary Artery Bypass Surgery: A Randomized Controlled Trial | postoperative 24 hours
  Postoperative visual pain score (VAS) monitoring, additional postoperative analgesic use, and patient satisfaction will be assessed by the pain nurse in the postoperative post-anesthesia care unit (PACU), where patients are routinely monitored for 24 hours.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Ankara
  - Ankara bilkent city hospital, Ankara, Çankaya 06530, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamed MA, Boules ML, Sobhy MM, Abdelhady MA. The Analgesic Efficacy of Ultrasound-Guided Bilateral Transversus Thoracic Muscle Plane Block After Open-Heart Surgeries: A Randomized Controlled Study. J Pain Res. 2022 Mar 5;15:675-682. doi: 10.2147/JPR.S355231. eCollection 2022. PMID 35281480
- [Background] Fang B, Wang Z, Huang X. Ultrasound-guided preoperative single-dose erector spinae plane block provides comparable analgesia to thoracic paravertebral block following thoracotomy: a single center randomized controlled double-blind study. Ann Transl Med. 2019 Apr;7(8):174. doi: 10.21037/atm.2019.03.53. PMID 31168455
- [Background] Abdallah NM, Bakeer AH, Youssef RB, Zaki HV, Abbas DN. Ultrasound-guided continuous serratus anterior plane block: dexmedetomidine as an adjunctive analgesic with levobupivacaine for post-thoracotomy pain. A prospective randomized controlled study. J Pain Res. 2019 Apr 30;12:1425-1431. doi: 10.2147/JPR.S195431. eCollection 2019. PMID 31118760
- [Background] Jannati M, Attar A. Analgesia and sedation post-coronary artery bypass graft surgery: a review of the literature. Ther Clin Risk Manag. 2019 Jun 20;15:773-781. doi: 10.2147/TCRM.S195267. eCollection 2019. PMID 31417264
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362
- [Background] Jack JM, McLellan E, Versyck B, Englesakis MF, Chin KJ. The role of serratus anterior plane and pectoral nerves blocks in cardiac surgery, thoracic surgery and trauma: a qualitative systematic review. Anaesthesia. 2020 Oct;75(10):1372-1385. doi: 10.1111/anae.15000. Epub 2020 Feb 16. PMID 32062870